CLINICAL TRIAL: NCT01200524
Title: A Study to Investigate the Analgesic Efficacy of AZD2423 Compared With Placebo After 28 Days Treatment in Patients With Posttraumatic Neuralgia..
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2600C00012
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Nerve Pain
Keywords: Analgesic effect
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD2423, 20mg (Experimental)
  Interventions: Drug: AZD2423
- AZD2423, 150 mg (Experimental)
  Interventions: Drug: AZD2423
- Placebo (Placebo Comparator): Tablet to match the 20 mg and 50 mg AZD2423 active tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2423 — 20 mg tablet
  Arms: AZD2423, 20mg
Drug: AZD2423 — 50 mg tablet
  Arms: AZD2423, 150 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A study to investigate the analgesic efficacy of AZD2423 compared with placebo after 28 days treatment in patients with posttraumatic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent form
* Males and female patients aged 18 to 80 years
* Patients with neuropathic pain due to peripheral nerve injury caused by trauma or surgery

Exclusion Criteria:

* Other paint that may confound assessment of neuropathic pain
* History of treatment failure with more than three adequate trials of treatment for neuropathic pain
* Central neuropathic pain conditions (caused by Central Nervous System injury/disease, eg. Stroke)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bror Jonzon, Study Director — AstraZeneca
Locations (25):
- Bulgaria (2):
  - Research Site, Pleven
  - Research Site, Sofia
- Denmark (2):
  - Research Site, Aalborg
  - Research Site, Odense
- France (4):
  - Research Site, Boulogne-Billancourt
  - Research Site, Clermont-Ferrand
  - Research Site, Nice
  - Research Site, Saint-Priest-en-Jarez
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Tychy
  - Research Site, Warsaw
- Russia (4):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Ufa
- Sweden (3):
  - Research Site, Falköping
  - Research Site, Kristianstad
  - Research Site, Stockholm
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Glasgow
  - Research Site, Manchester

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=205&filename=CSR-D2600C00012.pdf
- See also: CSR-D2600C00012.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=205&filename=CSR-D2600C00012.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 6th October 2010 and the last participant completed on 3rd April 2012. A total of 36 centres in France, Denmark, Poland, Russia, UK, Sweden and Bulgaria randomised 133 participants.
Pre-assignment Details: The study had an enrolment phase of up to 30 days (including wash-out period), a 28-day treatment phase, and a follow-up phase of 7-14 days. Participants were randomly assigned to blinded treatment in a 1:1:1 ratio either to AZD2423 20 mg, AZD2423 150 mg or placebo.
Groups:
- AZD2423, 150 mg: AZD2423 : 3x50 mg tablet once daily in the morning
- AZD2423, 20mg: AZD2423 : 1x20 mg tablet once daily in the morning
- Placebo: Tablet to match the 20 mg and 50 mg AZD2423 active tablet
  Placebo : Placebo
Period: Overall Study
Arm/Group | AZD2423, 150 mg | AZD2423, 20mg | Placebo
Started | 41 | 48 | 44
Completed | 39 | 47 | 40
Not Completed | 2 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Non availability of study nurse | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2423, 150 mg | AZD2423, 20mg | Placebo | Total
Number analyzed (Participants) | 41 | 48 | 44 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.9 (10.9) | 53.1 (10.9) | 55.1 (10.9) | 53.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 26 | 19 | 62
  Male | 24 | 22 | 25 | 71
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 41 | 47 | 44 | 132
  Black or African American | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Days 24-28 in Numerical Rating Scale (NRS) Average Pain Score.
Description: Last Observation Carried Forward (LOCF). Twice daily, the participants rated their Average Pain intensity during the past 12 hours on an Numerical Rating Scale (NRS) scale 0-10. 0= No pain, 10= Worst pain imaginable.
Time Frame: Baseline (mean of Day -5 to Day -1) to the mean of Day 24 to Day 28
Population: mITT analysis set including only those that had adequate NRS data at baseline and Days 24-28
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD2423, 150 mg | AZD2423, 20mg | Placebo
Number analyzed (Participants) | 41 | 47 | 43
Scores on a scale | -1.53 (1.67) | -1.54 (1.50) | -1.44 (1.59)

2. Secondary Outcome: Change From Baseline to Days 24-28 in Numerical Rating Scale (NRS) Worst Pain Score
Description: Last Observation Carried Forward (LOCF). Twice daily, the participants rated their Worst Pain intensity during the past 12 hours on an Numerical Rating Scale (NRS) 0-10; 0=No pain, 10=Worst pain imaginable.
Time Frame: Baseline (mean of Day -5 to Day -1) to the mean of Day 24 to Day 28
Population: mITT analysis set including only those that had adequate NRS data at baseline and Days 24-28
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD2423, 150 mg | AZD2423, 20mg | Placebo
Number analyzed (Participants) | 41 | 47 | 43
Scores on a scale | -1.8 (2.09) | -1.29 (1.5) | -1.4 (1.66)

3. Secondary Outcome: Number of Participants With at Least 30% Decrease From Baseline in Numerical Rating Scale (NRS) Average Pain Score at Day 28.
Description: LOCF- Last Observation Carried Forward. Numerical Rating Scale (NRS) Average Pain score reduction= (change from baseline at Day 28/baseline)*100. Responder=NRS Average Pain score reduction ≥30% (yes/no)
Time Frame: Baseline (mean of Day -5 to Day -1) to Day 28
Population: mITT analysis set
Measure: Number; unit: Participants
Arm/Group | AZD2423, 150 mg | AZD2423, 20mg | Placebo
Number analyzed (Participants) | 41 | 48 | 44
Participants | 17 | 15 | 17

4. Secondary Outcome: Number of Participants With at Least 50% Decrease From Baseline in Numerical RatingScale (NRS) Average Pain Score at Day 28.
Description: Last Observation Carried Forward (LOCF). Numerical Rating Scale (NRS) Average Pain score reduction=(change from baseline at Day 28/baseline)*100.
  Responder= NRS Average Pain score reduction ≥50% (yes/no)
Time Frame: Baseline (mean of Day -5 to Day -1) to Day 28
Population: mITT analysis set
Measure: Number; unit: Participants
Arm/Group | AZD2423, 150 mg | AZD2423, 20mg | Placebo
Number analyzed (Participants) | 41 | 48 | 44
Participants | 9 | 8 | 9

5. Secondary Outcome: Change From Baseline to Day 29 in Neuropathic Pain Symptom Inventory Scal (NPSI) Total Score.
Description: LOCF- Last Observation Carried Forward. At baseline and at end of treatment the participants filled in their Neuropathic Pain Symptom Inventory Scal (NPSI) pain symptom descriptors, recall period 24 hours. Each descriptor was rated on a NUmerical Rating Scale 0-10; 0=No (symptom), 10=Worst (symptom) imaginable. The NPSI Total Score was calculated as the sum of 10 of the NPSI descriptors. Higher total score is considered worse outcome.
Time Frame: Baseline (Day 1) to Day 29 (Visit 7)
Population: mITT analysis set including only those that had adequate NPSI data at baseline and Day 29
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD2423, 150 mg | AZD2423, 20mg | Placebo
Number analyzed (Participants) | 26 | 34 | 30
Scores on a scale | -16.58 (22.40) | -8.82 (18.11) | -9.8 (15.44)

ADVERSE EVENTS:
Arm/Group | AZD2423, 150 mg | AZD2423, 20mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/48 | 0/44
Other Adverse Events (participants affected / at risk) | 14/41 | 14/48 | 10/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2423, 150 mg (N=41) | AZD2423, 20mg (N=48) | Placebo (N=44)
Nausea (Gastrointestinal disorders) | 4 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1
Asthenia (General disorders) | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 5 | 4
Headache (Nervous system disorders) | 6 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement restricts the PI's rights to discuss or publish trial results after the trial is completed. No publication or presentation may include any of AZ's Confidential Information without AZ's prior written approval. AZ should have 60 days for review and can extend time until submission up to 90 days.